CLINICAL TRIAL: NCT03463681
Title: A Phase 2 Open Label Study of CaBozantinib in Patients With Advanced or Unresectable Renal cEll cArcinoma Pretreated With One immunochecKPOint INhibiTor (Anti PD1/PDL1): the BREAKPOINT Trial
Brief Title: A Study of CaBozantinib in Patients With Advanced or Unresectable Renal cEll cArcinoma
Acronym: BREAKPOINT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-000582-36
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): all subjects will recieve open label Cabozantinib 60 mg orally once daily
  Interventions: Drug: Cabometyx

INTERVENTIONS:
Drug: Cabometyx — cabozantinib 60 mg orally once daily
  Other Names: cabozantinib

SUMMARY:
This is an open label single arm, multicenter, phase II study designet To assess the progression free survival (PFS) of cabozantinib in patients pretreated with one immunocheckpoint inhibitor (CPI) in monotherapy or in combination

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. One previous anticancer treatment with a PD1/PDL1 inhibitor, as monotherapy or in combination with an angiogenesis inhibitor or anti CTLA 4, in both setting first line or adjuvant ( in this case patient having recurrence during the adjuvant treatment or within 6 months after therapy with PD1-PD-L1 therapy)
3. Age ≥18 years
4. Patients with histological diagnosis of predominant clear cells renal cell carcinoma
5. Measurable disease (as per RECIST 1.1 criteria) with documented radiological progression
6. Fertile women (<2 years after last menstruation) and men of childbearing potential must use effective methods of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgical sterilisation) during the study and for 4 months after the last dose of study treatment
7. All sites of disease including brain metastases (non symptomatic)
8. Karnofsky performance status ≥ 70%
9. Life expectancy greater than 3 months
10. The required values at baseline are as follows:

    * Absolute neutrophil count >1.5 x 109 /L,
    * Platelet count > 100 x 109 /L,
    * Haemoglobin > 9g/dl,
    * Total bilirubin < 1.5 upper limit of normal (ULN);
    * AST, ALT<2.5 ULN in patients without liver metastases, <5 ULN in patients with liver metastases;
    * serum creatinine < 2.0 mg/dl, amylase and lipase <1.5 ULN 11- Female subjects of childbearing potential must not be pregnant at screening

Exclusion Criteria:

1. Major surgical procedure within 28 days prior to study treatment start
2. Other malignancies within the last 5 years (other than curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix, meningiomas)
3. Clinically significant cardiovascular disease, for example cerebrovascular accidents (<6 months), myocardial infarction (<6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication
4. Recent (within the 30 days prior to randomisation) treatment with another investigational drug or participation in another investigational study
5. Symptomatic brain metastasis
6. History of other disease, metabolic dysfunction, physical examination finding or clinical laboratory finding giving reasonable suspicion of a disease condition that contraindicates use of an investigational drug or patient at high risk from treatment complications
7. PT or INR and PTT >1.5 times the Upper Normal Limit of the institution (patient who are being therapeutically anticoagulated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists).For patients on warfarin, close monitoring of at least weekly evaluations will be performed, until INR is stable based on a measurement at pre-dose, as defined by the local standard of care
8. Previous or concomitant radiotherapy in the lesion parameter of disease
9. Previous radiotherapy or other locoregional antitumoral treatment performed within 21 days before the study recruitment
10. Uncontrolled hypertension (>= 160 mmHg systolic and/or 90 mmHg diastolic) while receiving chronic medication
11. Inability to swallow tablets or capsules
12. Female subject who is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women
13. Known history of human immunodeficiency virus (HIV) infection, active hepatitis B, or active hepatitis C.
14. Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
progression free survival (PFS) | 28 month
  To assess the progression free survival (PFS) of cabozantinib in patients pretreated with one immunocheckpoint inhibitor (CPI) in monotherapy or in combination

SECONDARY OUTCOMES:
overall survival (OS) | 28 month
  To assess the overall survival (OS)
objective response rates (ORR) | 28 month
  the efficacy based on objective response rates (ORR) according to RECIST 1:1 criteria
safety: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 28 month
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Procopio, MD, Principal Investigator — Fondazione IRCCS ISTITUTO NAZIONALE TUMORI
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Derosa L, Rouche JA, Colomba E et al. Efficacy of cabozantinib after PD1/PDL1 checkpoint inhibitors in metastatic renal cell carcinoma (mRCC): the gustave Roussy experience. Ann of Onc vol 28, sep 2017
- [Background] Shah A, Lemke E, Gao J et al, Outcomes of patients with metastatic clear cell renal cell carcinoma treated with second line vascular endothelial growth factor receptor tyrosine kinase inhibitors after first line immune checkpoint inhibitors; Genitourinary Cancer Symposium 2018, abstract 682.
- [Background] Ref: Brookmeyer, R and Crowley, JJ (1982): A confidence interval for the median survival time. Biometrics 38:29-41
- [Result] Choueiri TK, Escudier B, Powles T, Mainwaring PN, Rini BI, Donskov F, Hammers H, Hutson TE, Lee JL, Peltola K, Roth BJ, Bjarnason GA, Geczi L, Keam B, Maroto P, Heng DY, Schmidinger M, Kantoff PW, Borgman-Hagey A, Hessel C, Scheffold C, Schwab GM, Tannir NM, Motzer RJ; METEOR Investigators. Cabozantinib versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1814-23. doi: 10.1056/NEJMoa1510016. Epub 2015 Sep 25. PMID 26406150
- [Result] Choueiri TK, Escudier B, Powles T, Tannir NM, Mainwaring PN, Rini BI, Hammers HJ, Donskov F, Roth BJ, Peltola K, Lee JL, Heng DYC, Schmidinger M, Agarwal N, Sternberg CN, McDermott DF, Aftab DT, Hessel C, Scheffold C, Schwab G, Hutson TE, Pal S, Motzer RJ; METEOR investigators. Cabozantinib versus everolimus in advanced renal cell carcinoma (METEOR): final results from a randomised, open-label, phase 3 trial. Lancet Oncol. 2016 Jul;17(7):917-927. doi: 10.1016/S1470-2045(16)30107-3. Epub 2016 Jun 5. PMID 27279544
- [Result] Choueiri TK, Halabi S, Sanford BL, Hahn O, Michaelson MD, Walsh MK, Feldman DR, Olencki T, Picus J, Small EJ, Dakhil S, George DJ, Morris MJ. Cabozantinib Versus Sunitinib As Initial Targeted Therapy for Patients With Metastatic Renal Cell Carcinoma of Poor or Intermediate Risk: The Alliance A031203 CABOSUN Trial. J Clin Oncol. 2017 Feb 20;35(6):591-597. doi: 10.1200/JCO.2016.70.7398. Epub 2016 Nov 14. PMID 28199818
- [Result] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Result] Cella D, Escudier B, Tannir NM, Powles T, Donskov F, Peltola K, Schmidinger M, Heng DYC, Mainwaring PN, Hammers HJ, Lee JL, Roth BJ, Marteau F, Williams P, Baer J, Mangeshkar M, Scheffold C, Hutson TE, Pal S, Motzer RJ, Choueiri TK. Quality of Life Outcomes for Cabozantinib Versus Everolimus in Patients With Metastatic Renal Cell Carcinoma: METEOR Phase III Randomized Trial. J Clin Oncol. 2018 Mar 10;36(8):757-764. doi: 10.1200/JCO.2017.75.2170. Epub 2018 Jan 29. PMID 29377755
- [Result] Motzer RJ, Hutson TE, Cella D, Reeves J, Hawkins R, Guo J, Nathan P, Staehler M, de Souza P, Merchan JR, Boleti E, Fife K, Jin J, Jones R, Uemura H, De Giorgi U, Harmenberg U, Wang J, Sternberg CN, Deen K, McCann L, Hackshaw MD, Crescenzo R, Pandite LN, Choueiri TK. Pazopanib versus sunitinib in metastatic renal-cell carcinoma. N Engl J Med. 2013 Aug 22;369(8):722-31. doi: 10.1056/NEJMoa1303989. PMID 23964934
- [Derived] Procopio G, Claps M, Pircher C, Porcu L, Sepe P, Guadalupi V, De Giorgi U, Bimbatti D, Nole F, Carrozza F, Buti S, Iacovelli R, Ciccarese C, Masini C, Baldessari C, Doni L, Cusmai A, Gernone A, Scagliarini S, Pignata S, de Braud F, Verzoni E. A multicenter phase 2 single arm study of cabozantinib in patients with advanced or unresectable renal cell carcinoma pre-treated with one immune-checkpoint inhibitor: The BREAKPOINT trial (Meet-Uro trial 03). Tumori. 2023 Feb;109(1):129-137. doi: 10.1177/03008916221138881. Epub 2022 Nov 29. PMID 36447337